CLINICAL TRIAL: NCT01111721
Title: Adapting Project SAFE: Reducing STD/HIV Risk in Women Prisoners
Brief Title: Project POWER, Adapting Project SAFE: Reducing STD/HIV Risk in Women Prisoners
Acronym: POWER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Catherine Fogel, PhD, Professor-Principle Investigator, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 09-1433; 5UR6PS000670 (NIH)
Record Dates: First submitted 2010-04-05; First posted 2010-04-28 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: HIV Infections
Keywords: Sexually Transmitted Diseases; HIV Infections; Genital Diseases, Female; Acquired Immunodeficiency Syndrome; Risk Reduction Behavior; HIV prevention
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases; Genital Diseases, Female; Acquired Immunodeficiency Syndrome; Risk Reduction Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Project POWER Intervention Group (Experimental): Intervention group participants will attend the Project POWER intervention sessions, complete a pre-intervention assessment and participate in 3, 6, and 12 month follow-up interviews when they will be asked to provide urine specimens for STI testing. The intervention consists of eight bi-weekly, 1.5 hour sessions. Intervention group participants will also attend one booster group session four weeks after the intervention before being released. Intervention participants will receive booster phone calls from a nurse-interventionist at 2, 6, and 10 weeks after release from prison. Booster phone calls will reinforce intervention content and support participant efforts to reduce risky sex behaviors and make healthy choices.
  Interventions: Behavioral: Project POWER HIV Risk-reduction Intervention
- NC DOC Standard of Care for STIs (Active Comparator): Control group participants will receive the North Carolina Department of Correction standard of care for Sexually Transmitted Infections, complete one interview in prison and participate in 3, 6, and 12 month follow up interviews when they will be asked to provide urine specimens for STI testing.
  Interventions: Behavioral: NC DOC Standard of Care for STIs

INTERVENTIONS:
Behavioral: Project POWER HIV Risk-reduction Intervention — Nine session group-based behavioral intervention for incarcerated female adults.
  Arms: Project POWER Intervention Group
Behavioral: NC DOC Standard of Care for STIs — Standard North Carolina Department of Correction intake STI testing and counseling.
  Arms: NC DOC Standard of Care for STIs

SUMMARY:
Project POWER will test the efficacy of a multi-session HIV Prevention program, adapted from an existing program (Project SAFE), for incarcerated women in the rural South.

DETAILED DESCRIPTION:
Incarcerated women have a disproportionately high risk for both Sexually Transmitted Infections (STIs) and Human Immunodeficiency Virus (HIV)/Acquired Immune Deficiency Syndrome (AIDS)and the prevalence of HIV and STIs are higher among women than men prisoners. More than half of the HIV/AIDS cases reported by State and Federal prisons in 2005 were in the South. The second highest regional burden for HIV among women released from correction facilities is in the South.

Working in collaboration, the staff of the North Carolina Department of Correction (NCDOC) and faculty at the University of North Carolina at Chapel Hill School of Nursing (SON), School of Medicine (SOM), Center for AIDS Research (CFAR) and the School of Social Work (SSW) will systematically adapt and test the efficacy of Project SAFE, an existing evidence-based intervention (EBI), to increase protective behaviors, reduce high-risk behaviors, and prevent STIs in HIV-negative incarcerated women in the Southern United States.

Using Centers for Disease Control and Prevention (CDC) guidelines for adaptation (McKleroy, Galbraith, Cummings et al. 2006), we will:

1. Assess the fit between intervention delivery and the needs and resources of the NCDOC and the fit between intervention materials and the behavioral, social, and contextual conditions of incarcerated women's lives following release from prison that may contribute to continuing sexual risk behavior and explore their ideas regarding ways to prevent STI/HIV with the intent of strengthening the approach to sexual risk reduction.
2. Adapt and tailor the Project SAFE behavioral risk reduction intervention for women prisoners in the rural Southeastern U.S. who are HIV-negative and have sex with men.
3. Pilot the adapted Project SAFE intervention.
4. Test the adapted Project SAFE risk-reduction intervention with incarcerated women to determine its efficacy in decreasing risk for non-viral STI infections (Chlamydia, trichomoniasis or gonorrhea), decreasing sexual risk behaviors and increasing risk reduction practices after release. We will also determine whether participants maintain these changes over time.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* Ability to provide verbal and written consent
* A plan to reside in North Carolina after release from prison and for the length of the study
* Sentence length of 12 months or less with less than 6 months to serve
* Anticipated sexual activity with a man
* Access to a telephone after release
* HIV negative status

Exclusion Criteria:

* Under age 18
* Unable to speak and read English
* Plan to live somewhere other than in North Carolina
* Sentence lengths of more than 12 months, or 12 months but with more than 6 months to serve
* Individuals who exhibit signs of acute intoxication or appear to be under the influence of drugs, or exhibit an inability to focus or understand explanations, or exhibit symptoms of acute psychosis
* No access to a telephone after release
* HIV-positive status (determined by self-report)
* Participation in the pilot phase

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 598 (Actual)
Dates: Start 2009-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
STI Infection Rate | 12 months after release from prison

SECONDARY OUTCOMES:
Number of unprotected sex acts as a measure of enacting sexual protective practices. | 12 months after release from prison.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine I. Fogel, PhD, Principal Investigator — School of Nursing, The University of North Carolina at Chapel Hill
Locations (2):
- United States (2):
  - North Carolina Correctional Institution for Women, Raleigh, North Carolina
  - Fountain Correctional Center for Women, Rocky Mount, North Carolina

REFERENCES:
- [Derived] Herbst JH, Branscomb-Burgess O, Gelaude DJ, Seth P, Parker S, Fogel CI. Risk Profiles of Women Experiencing Initial and Repeat Incarcerations: Implications for Prevention Programs. AIDS Educ Prev. 2016 Aug;28(4):299-311. doi: 10.1521/aeap.2016.28.4.299. PMID 27427925